CLINICAL TRIAL: NCT00886366
Title: A Randomised, Single-Blind, Placebo-Controlled, Single-Centre, Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food Interaction After Single Ascending Oral Doses of AZD6714 in Healthy Male Volunteers and Male Type II Diabetic Patients
Brief Title: Single Ascending Dose Study With Healthy Male Volunteers and Type II Diabetic Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part A reached a predefined stopping criteria. Relevant doses for part B could not be established based on A and subsequently study was stopped.
Sponsor: AstraZeneca (Industry)
Responsible Party: Klas Malmberg, MD, PhD, Prof. Medical Science Director, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: D1920C00001
Record Dates: First submitted 2009-04-17; First posted 2009-04-22 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Type 2 Diabetes
Keywords: Type II Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- 1 (Experimental): AZD6714 in 8 increasing oral single doses a-h given to 8 groups (3 on active and 1 on placebo in each group)
  Interventions: Drug: AZD6714; Drug: Placebo
- 2 (Experimental): 2 oral single doses d and g suspensions of AZD6714 given to 2 groups (3+1) together with food
  Interventions: Drug: Placebo; Drug: AZD6714
- 3 (Experimental): Two increasing oral doses of AZD6714 and one placebo given to 2 groups with 3 type 2 diabetic patients.
  Interventions: Drug: Placebo; Drug: AZD6714

INTERVENTIONS:
Drug: AZD6714 — Oral single doses a-h suspension
  Arms: 1
Drug: Placebo — Oral single doses suspension
Drug: AZD6714 — Oral single doses a-d suspension
  Arms: 3
Drug: AZD6714 — Oral single doses d and g suspension
  Arms: 2

SUMMARY:
The purpose of this study is to assess safety and tolerability of AZD6714 after single ascending oral doses in healthy male subjects and type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Part A,Healthy male subjects, aged between ≥20 and ≤40 years.
* Part B,Male T2DM patients, aged between ≥20 and ≤65 years. Treatment with metformin as single therapy for T2DM for at least 30 days prior to enrollment

Exclusion Criteria:

* Part A,Clin sign illness or clin relevant trauma, as judged by the investigator, within 2 weeks before the first administration of the IP.
* Part A Clin sign abnormalities in clinical chemistry, haematology, or urinalysis results as judged by the investigator
* Part B, History of ischemic heart disease, symptomatic heart failure, stroke, transitory ischemic attack or symptomatic peripheral vascular disease.
* Any clinically significant abnormality identified on physical examination, laboratory tests or ECG, which in the judgment of the investigator would compromise the patient's safety or successful participation.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety variables (AE, BP, pulse, plasma glucose, laboratory variables and ECG) | AEs will be collected during the whole study period (1-3 months). The other variables will be measured repeatedly during 24 hours on the study day sessions

SECONDARY OUTCOMES:
Pharmacokinetic variables | Blood samples taken repeatedly during 24 hours on study day sessions.
Pharmacodynamic variables (P-Glucose, S-Insulin and C-peptide) | Blood samples taken repeatedly during 24 hours on study day sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Study Director — AstraZeneca R&D Mölndal; Marianne Hartford, Principal Investigator — CPU Sahlgrenska University Hospital
Locations (1):
- Research Site, Gothenburg, Sweden